CLINICAL TRIAL: NCT03506412
Title: A Proof of Concept Study to Determine the Efficacy of Entresto™ in HFpEF Based on Circulating Neprilysin Levels: The Circulating NEP and NEP Inhibition (CNEPi) Study
Brief Title: Circulating NEP and NEP Inhibition Study in Heart Failure With Preserved Ejection Fraction
Acronym: CNEPi
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Naveen L. Pereira, Professor of Medicine, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-000044; R21AG053512 (NIH)
Record Dates: First submitted 2018-04-11; First posted 2018-04-24 (Actual); Results first posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: Heart Failure; HFpEF; Entresto™; Neprilysin; Diastolic Heart Failure
MeSH Terms: conditions — Heart Failure; Heart Failure, Diastolic | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Intervention Model Description: Entresto™ will be administered to subjects with high and low circulating neprilysin (NEP) levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low Serum Neprilysin (sNEP) levels (Experimental): Subjects with baseline sNEP levels less than or equal to 0.9 ng/ml
  Interventions: Drug: Entresto™ 49Mg-51 mg tablet
- High Serum Neprilysin (sNEP) levels (Experimental): Subjects with baseline sNEP greater than or equal to 0.9 ng/ml
  Interventions: Drug: Entresto™ 49Mg-51 mg tablet

INTERVENTIONS:
Drug: Entresto™ 49Mg-51 mg tablet — Entresto™ 49Mg-51 mg will be given twice daily orally for 5 weeks

SUMMARY:
To determine biomarker responses to Entresto™in patients with Heart Failure with preserved Ejection Fraction (HFpEF) and who have high or low serum neprilysin (NEP) levels.

DETAILED DESCRIPTION:
This is a proof of concept single arm study in which 40 subjects with HFpEF will be assigned to Entresto™ 49/51 mg (sacubitril/valsartan) twice-daily for a total duration of up to 5 weeks of treatment. Blood will be drawn prior to and at completion of treatment. The primary endpoint measured is change in biomarkers with Entresto™ administration that reflect NEP activity and myocardial stress (NT pro-ANP, -BNP, -CNP) and drug action (cGMP). This endpoint has been well validated as a measure of Entresto™ drug response.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 50 years
2. LVEF ≥ 45% assessed by echocardiography, nuclear scan, MRI or left ventriculogram within the past 24 months
3. Current New York Heart Association (NYHA) class 2-4 symptoms of heart failure (HF)
4. Stable medical therapy for 30 days as defined by:

   1. No addition or removal of ACE, ARB, beta-blockers, calcium channel blockers (CCBs) or aldosterone antagonists
   2. No change in dosage of ACE, ARBs, beta-blockers, CCBs or aldosterone antagonists of more than 100%
5. One of the following within the last 24 months

   1. Previous hospitalization for HF with radiographic evidence of pulmonary congestion (pulmonary venous hypertension, vascular congestion, interstitial edema, pleural effusion) or
   2. Catheterization documented elevated filling pressures at rest (LVEDP≥15 or PCWP≥20) or with exercise (PCWP≥25) or
   3. Elevated NT-proBNP (> 400 pg/ml) or BNP (> 200 pg/ml) or
   4. Echo evidence of diastolic dysfunction / elevated filling pressures (at least two)

   i. E/A > 1.5 + decrease in E/A of > 0.5 with valsalva

ii. Deceleration time ≤ 140 ms

iii. Pulmonary vein velocity in systole < diastole (PVs<PVd) (sinus rhythm)

iv. E/e'≥15

v. Left atrial enlargement (≥ moderate)

vi. Pulmonary artery systolic pressure > 40 mmHg

vii. Evidence of left ventricular hypertrophy

1. LV mass/BSA ≥ 96 (♀) or ≥ 116 (♂) g/m2
2. Relative wall thickness ≥ 0.43 (♂ or ♀) [(IVS+PW)/LVEDD]
3. Posterior wall thickness ≥ 0.9 (♀) or 1.0 (♂) cm

Exclusion Criteria

1. History of hypersensitivity or allergy to ACE inhibitors (ACEIs), ARBs, or NEP inhibitors
2. Known history of angioedema
3. Previous LVEF < 40% at any time
4. Systolic blood pressure < 100 mmHg or > 180 mmHg
5. Current acute decompensated HF (exacerbation of chronic HF manifested by signs and symptoms that may require intravenous therapy)
6. Unstable angina, myocardial infarction, stroke, transient ischemic attack, or cardiovascular surgery or urgent percutaneous coronary intervention (PCI) within 3 months of screening or elective PCI within 30 days of entry
7. Significant valvular stenosis or regurgitation (greater than moderate in severity), hypertrophic, restrictive or obstructive cardiomyopathy including amyloidosis, constrictive pericarditis, primary pulmonary hypertension, or biopsy proven active myocarditis
8. Severe congenital heart disease
9. History of heart transplant or with LV assist device
10. Evidence of severe hepatic disease as determined by any one of the following: history of hepatic encephalopathy, history of esophageal varices, or history of porto-caval shunt.
11. Glomerular filtration rate < 20 ml/min/1.73 m2 on most recent clinical laboratories*
12. Serum potassium of > 5.5 mEq/dL on most recent clinical laboratories*
13. Concomitant use of aliskiren in patients with diabetes
14. Currently receiving an investigational drug
15. Inability to comply with planned study procedures
16. Female subject who is pregnant or breastfeeding

    * Performed within 90 days of enrollment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naveen L Pereira, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total of 40 subject enrolled. Enrolled subjects were assigned to an arm based on their Baseline serum Neprilysin (sNEP) levels. Baseline sNEP levels were only available for 37 subjects. Data not collected for 3 subjects.
Groups:
- Low Serum Neprilysin (sNEP) Levels: Subjects with baseline sNEP levels less than or equal to 0.9 ng/ml
  Entresto™ 49Mg-51 mg tablet: Entresto™ 49 Mg-51 mg will be given twice daily orally for 5 weeks
- High Serum Neprilysin (sNEP) Levels: Subjects with baseline sNEP greater than or equal to 0.9 ng/ml
  Entresto™ 49Mg-51 mg tablet: Entresto™ 49 Mg-51 mg will be given twice daily orally for 5 weeks
Period: Overall Study
Arm/Group | Low Serum Neprilysin (sNEP) Levels | High Serum Neprilysin (sNEP) Levels
Started | 18 | 19
Completed | 18 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total of 40 subject enrolled. Enrolled subjects were assigned to an arm based on their Baseline serum Neprilysin (sNEP) levels. Baseline sNEP levels were only available for 37 subjects. Data not collected for 3 subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Serum Neprilysin (sNEP) Levels | High Serum Neprilysin (sNEP) Levels | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 77.0 [72.0 to 86.0] | 74.0 [63.0 to 78.0] | 76 [71 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 8 | 12 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma N-terminal Proatrial Natriuretic Peptide (NT proANP)
Description: Change in plasma NT pro-ANP value levels as measured in pg/mL. NT-pro ANP means N-terminal polypeptide of ANP (atrial natriuretic peptide) precursor. Natriuretic peptides are substances made by the heart. Elevated levels can mean the heart isn't pumping as much blood the body needs.
Time Frame: baseline, 5 weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Low Serum Neprilysin (sNEP) Levels | High Serum Neprilysin (sNEP) Levels
Number analyzed (Participants) | 18 | 19
pg/mL | 47.4 [-4.6 to 129.9] | 46.4 [6.4 to 139.5]

2. Primary Outcome: Change in Plasma N-terminal Pro B-type Natriuretic Peptide (NT-proBNP)
Description: Change in plasma NT pro-ANP value levels as measured in pg/mL. Natriuretic peptides are substances made by the heart. Two main types of these substances are brain natriuretic peptide (BNP) and N-terminal pro b-type natriuretic peptide (NT-proBNP). Elevated levels can mean the heart isn't pumping as much blood the body needs.
Time Frame: baseline, 5 weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Low Serum Neprilysin (sNEP) Levels | High Serum Neprilysin (sNEP) Levels
Number analyzed (Participants) | 18 | 19
pg/mL | -11.5 [-50.0 to 66.0] | 45.0 [-16.0 to 107.0]

3. Primary Outcome: Change in Plasma N-terminal Brain Natriuretic Peptide (BNP)
Description: Change in plasma BNP biomarker value levels as measured in pg/mL. Brain natriuretic peptide is a hormone secreted by cardiomyocytes in the heart ventricles in response to stretching caused by increased ventricular blood volume. Elevated levels can mean the heart isn't pumping as much blood the body needs.
Time Frame: baseline, 5 weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Low Serum Neprilysin (sNEP) Levels | High Serum Neprilysin (sNEP) Levels
Number analyzed (Participants) | 18 | 19
pg/mL | -301.5 [-684.0 to -20.0] | -100.0 [-405.0 to 69.0]

4. Primary Outcome: Change in Plasma Cyclic Guanine Monophosphate (cGMP)
Description: Change in Plasma cGMP biomarker value levels as measured in nmol/L. Cyclic guanosine monophosphate is a cyclic nucleotide derived from guanosine triphosphate. cGMP acts as a second messenger to tissue and cellular responses.
Time Frame: baseline, 5 weeks
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | Low Serum Neprilysin (sNEP) Levels | High Serum Neprilysin (sNEP) Levels
Number analyzed (Participants) | 18 | 19
nmol/L | 4.2 [2.4 to 8.5] | 1.0 [-0.9 to 6.3]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 5 weeks
Arm/Group | Low Serum Neprilysin (sNEP) Levels | High Serum Neprilysin (sNEP) Levels
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 0/18 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/12/NCT03506412/Prot_SAP_000.pdf